CLINICAL TRIAL: NCT00281424
Title: Increasing Walking Following Completion of Cardiac Rehabilitation
Brief Title: Increasing Walking Following Cardiac Rehabilitation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-080105
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Diseases; Walking
Keywords: exercise adherence; cardiac patients; walking
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): no pedometer
- pedometer (Experimental): given pedometer
  Interventions: Device: pedometer

INTERVENTIONS:
Device: pedometer — gave pedometer and info
  Arms: pedometer

SUMMARY:
The purpose of the project was to test the widely endorsed assumption that pedometers produce or encourage more physical activity participation in the form of walking. The investigators hypothesized that pedometers would not increase the amount of walking cardiac patients participated in after their cardiac rehabilitation program compared to patients without pedometers.

DETAILED DESCRIPTION:
As evidenced by the media attention given to pedometers and recent physical activity promotional efforts focused on pedometers, people seem to think that owning a pedometer will influence activity levels.

However, an examination of a few social cognitive theories produces no theoretical rationale that would support any sustained positive influence of pedometers in the absence of some other conditional factor, such as a behavioural goal or a social support system. We believe that once people determine how many steps their usual routes and daily activity typically amounts to, that the pedometer will no longer be used. We based our contentions on two theories: self efficacy theory (Bandura, 1986;1997) and self-determination theory (Deci & Ryan, 2000).

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the Northern Alberta Cardiac Rehabilitation Program
* Patients who are willing to participate
* Are able to read English
* Patients who are able to walk at 2.0 mph based on their exercise stress test results

Exclusion Criteria:

* patients unable to walk or walking contra-indicated
* unwilling
* do not read English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Physical activity behaviour | months

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Rodgers, PhD, Principal Investigator — University of Alberta
Locations (1):
- Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No